CLINICAL TRIAL: NCT07271121
Title: A Phase II Study of CART Cell (MB-CART19.1) in Patients With Relapsed or Refractory CD19 Positive NHL
Brief Title: Study of CART Cell (MB-CART19.1) in Patients With Relapsed or Refractory CD19 Positive NHL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24 KHCC 192
Record Dates: First submitted 2025-11-24; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Non-Hodgkin Lymphoma Refractory/ Relapsed
Keywords: Non-Hodgkin Lymphoma Refractory/ Relapsed; MB-CART-19.1

STUDY DESIGN:
Intervention Model Description: This is a prospective single center, open label, non-randomized, single arm, single dose, optimal 2-stage Simon design, and Phase II clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MB-CART-19.1 (Experimental): One dose of fresh MB-CART-19.1 at dose level 1- 3x10^6/kg ABW for patients. The leukapheresed product will be used for the individual manufacturing of MB-CART19.1 by using the automated closed CliniMACS Prodigy System
  Interventions: Other: MB-CART-19.1

INTERVENTIONS:
Other: MB-CART-19.1 — The leukapheresed product will be used for the individual manufacturing of MB-CART19.1 by using the automated closed CliniMACS Prodigy System. CD4+ and CD8+ T-cells will be selected, enriched and activated, followed by lentivirus-based transduction with the CD19 CAR construct. Then the MB-CART19.1 transduced T cells will be expanded and finally formulated.

SUMMARY:
This is a Prospective Single Center, open label, Non-randomized, Single Arm, Single Dose, Phase II Clinical Trial. Adult patients >18-year-old with CD19+ Non-Hodgkin lymphoma are eligible for the study if they meet eligibility criteria. Patients will receive a fresh single dose of MB-CART-19.1 and will be followed for 12 months and evaluated for efficacy and safety.

DETAILED DESCRIPTION:
This is a prospective single center, open label, non-randomized, single arm, single dose, optimal 2-stage Simon design, and Phase II clinical trial. The trial includes Adult patients > 18-year-old and up to 75 years old, with CD19+ non-Hodgkin lymphoma including diffuse Large B-cell Lymphoma, primary mediastinal B-cell lymphoma and relapsed refractory follicular lymphoma.

Single infusion of freshly prepared MB-CART19.1 cells manufactured according to Miltinyi Biotec product manufacturing guidelines and good manufacturing product (GMP) of KHCC manufacturing standard operating procedures (SOPs).

The patients will receive one infusion of the MB-CART19.1 product in infusion solution at a final volume adapted to the patients' weight, over a time of approx. 5-20 minutes (intravenous infusion via a large peripheral vein or central line).

The objective of this trial is to assess the efficacy and safety of ex vivo generated MB-CART19.1 in adult patients with relapsed or refractory CD19 positive Non-Hodgkin lymphoma including diffuse Large B-cell Lymphoma, primary mediastinal B-cell lymphoma and relapsed refractory follicular lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients with a diagnosis of aggressive NHL:

   1. Patients after progression on at least one standard chemotherapy and one salvage regimen or
   2. Patients considered for alloSCT but are found ineligible or
   3. Patients who have relapsed post alloSCT at least 100 days post-transplant, with no evidence of active GVHD, and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.
2. Patients with CNS disease (excluding isolated CNS lymphoma) are eligible only if disease has been successfully cleared at the time of inclusion.
3. CD19 expression must be detected on the malignant cells by flow cytometry or immunohistochemistry
4. Age > 18 year up to 75 years old (if deemed fit by treating investigator);
5. Baseline absolute CD3+ T cell count by FACS ≥100/µl;
6. ECOG performance score of 0-2 at screening;
7. No active Hepatitis B, Hepatitis C, HIV I/II
8. No childbearing potential or negative pregnancy test at screening within 7 days from starting lymphodepletion chemotherapy and before bridging chemotherapy in women with childbearing potential;
9. Signed and dated informed consent, before conduct of any trial-specific procedure.

Exclusion Criteria:

1. Residual CNS disease
2. Current autoimmune disease, or history of autoimmune disease with potential CNS involvement;
3. Active clinically significant CNS dysfunction (including but not limited to uncontrolled seizure disorders, cerebrovascular ischemia or hemorrhage, dementia, paralysis)
4. History of an additional malignancy other than non-melanoma skin cancer or carcinoma in situ unless disease free for ≥3 years;
5. Pulmonary function: Patients with pre-existing severe lung disease or DLCO of less than 50% or active pulmonary infiltrates on imaging studies.
6. Cardiac function: left ventricular ejection faction <50% by echocardiogram,
7. Renal function: Creatinine clearance <50 mL/min/1.73 m2, by Cockcroft-Gault formula (Cockcroft and Gault 1976) for patients ≥18 years.
8. Liver function: patients with serum bilirubin ≥3 times upper limit of or AST or ALT > 5 times upper limit of normal, unless due to lymphoma liver infiltration in the estimation of the investigator.
9. Rapidly progressive disease that in the estimation of the investigator would compromise ability to complete study therapy;
10. Pregnant or breast-feeding females
11. Medications: systemic chemotherapies, corticosteroids with the exception of physiologic replacement dosing, Fludarabine/clofarabine or immunosuppressive (Calcineurin inhibitors) drugs and antibodies or investigational drugs or donor lymphocyte transfusions or radiation therapy within 30 days prior to apheresis, and rituximab within 2 weeks with the exception of Intrathecal chemotherapy is allowed prior to treatment, but should be discontinued 10 days prior to-CART19 infusion to limit the risk of neurotoxicities;
12. Patients of child-bearing or fathering potential not willing to practice an effective form of birth control from the time of enrollment and for three months after dosing of the CARTs;
13. Concurrent participation in another interventional trial that could interact with this trial, e.g. CAR T trials.
14. Other investigational treatment within 4 weeks before CARTs infusion;
15. Cerebral dysfunction, legal incapacity of adult patients;
16. Committal to an institution on judicial or official order.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate | on week 4 and at month 3 in patients not achieving CR on week 4
  ORR in NHL patients defined as the rate of overall response (CR or PR)

SECONDARY OUTCOMES:
Safety and toxicity | From enrolment to the end of follow up at one year
  Safety and toxicity of MB-CART19.1, Overall incidence and severity of adverse events
CRS | From enrolment to the end of follow up at one year
  The incidence rate of CRS
Disease-free survival | at 1 year after receiving study treatment
  Disease-free at 1 year after MB-CART 19.1 in patients not receiving alloHCT
Duration of response | From enrolment to end of follow up at one year
  Duration of response
ICANS | From enrolment to the end of follow up at one year
  The incidence rate of ICANS
relapse rate | From enrolment to the end of follow up at one year
  relapse rate
time to relapse | From enrolment to the end of follow up at one year
  time to relapse
overall survival | at 1 year after receiving study treatment
  overall survival at 1 year after MB-CART 19.1 in patients not receiving alloHCT

CONTACTS AND LOCATIONS:
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
to maintain privacy and confidentiality of personal data